CLINICAL TRIAL: NCT01950520
Title: The Mechanism of Human Non-Shivering Thermogenesis and Basal Metabolic Rate
Brief Title: Study of Human Non-Shivering Thermogenesis and Basal Metabolic Rate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 130200; 13-DK-0200
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-06-11

CONDITIONS: Healthy Volunteers
Keywords: Adipose Tissue; Adult; Resting Energy Expenditure; RESPIRATORY QUOTIENT; BASAL METABOLIC RATE
MeSH Terms: interventions — Propranolol; Pindolol; Dantrolene; Magnesium Sulfate; Caffeine; Qsymia; Topiramate; Phentermine; Naltrexone; mirabegron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Chamber temperature will be block randomized with low temperature and 27°C (Cohort 1 only)
  Within each block, the following five interventions will be repeated:
  Propranolol: Propanolol 160mg, oral, by mouth (Cohort 1 only)
  Pindolol: Pindolol 20mg, oral, by mouth (Cohort 1 only)
  Dantrolene: Dantrolene 100mg, oral, by mouth (Cohort 1 only)
  Magnesium Sulfate: Magnesium Sulfate, infusion, 50 mg/kg bolus followed by maintenance infusion at 2g/h (Cohort 1 only)
  Placebo Cohort 1: Placebo, oral, by mouth (Cohort 1 only)
  Interventions: Drug: Propranolol; Drug: Pindolol; Drug: Dantrolene; Drug: Magnesium Sulfate; Drug: Placebo Cohort 1
- Cohort 2 (Experimental): Interventions, in random order, will be administered during one of the six one-day stays
  Caffeine: Caffeine 200mg, oral, by mouth (Cohort 2 only)
  Qsymia: Qsymia (topiramate 92mg CR, phentermine 15mg PO), oral, by mouth (Cohort 2 only)
  Topiramate: Topiramate 200mg, oral, by mouth (Cohort 2 only)
  Phentermine: Phentermine 37.5mg, oral, by mouth (Cohort 2 only)
  Naltrexone: Naltrexone 100mg, oral, by mouth (Cohort 2 only)
  Placebo Cohort 2: Placebo, oral, by mouth (Cohort 2 only)
  Interventions: Drug: Caffeine; Drug: Qsymia; Drug: Topiramate; Behavioral: Phentermine; Drug: Naltrexone; Drug: Placebo Cohort 2
- Cohort 3 (Experimental): Interventions, in random order, will be administered during one of the four overnight inpatient stays
  Mirabegron 50mg: Mirabegron 50mg, oral, by mouth (Cohort 3 only)
  Mirabegron 200mg: Mirabegron 200mg, oral, by mouth (Cohort 3 only)
  Placebo for Mirabegron: Placebo for Mirabegron, oral, by mouth (Cohort 3 only)
  Interventions: Drug: Mirabegron 50mg; Drug: Mirabegron 200mg; Drug: Placebo for Mirabegron

INTERVENTIONS:
Drug: Propranolol — Propanolol 160mg, oral, by mouth (Cohort 1 only)
  Arms: Cohort 1
Drug: Pindolol — Pindolol 20mg, oral, by mouth (Cohort 1 only)
  Arms: Cohort 1
Drug: Dantrolene — Dantrolene 100mg, oral, by mouth (Cohort 1 only)
  Arms: Cohort 1
Drug: Magnesium Sulfate — Magnesium Sulfate, infusion, 50 mg/kg bolus followed by maintenance infusion at 2g/h (Cohort 1 only)
  Arms: Cohort 1
Drug: Caffeine — Caffeine 200mg, oral, by mouth (Cohort 2 only)
  Arms: Cohort 2
Drug: Qsymia — Qsymia (topiramate 92mg CR, phentermine 15mg PO), oral, by mouth (Cohort 2 only)
  Arms: Cohort 2
Drug: Topiramate — Topiramate 200mg, oral, by mouth (Cohort 2 only)
  Arms: Cohort 2
Behavioral: Phentermine — Phentermine 37.5mg, oral, by mouth (Cohort 2 only)
  Arms: Cohort 2
Drug: Naltrexone — Naltrexone 100mg, oral, by mouth (Cohort 2 only)
  Arms: Cohort 2
Drug: Mirabegron 50mg — Mirabegron 50mg, oral, by mouth (Cohort 3 only)
  Arms: Cohort 3
Drug: Mirabegron 200mg — Mirabegron 200mg, oral, by mouth (Cohort 3 only)
  Arms: Cohort 3
Drug: Placebo Cohort 1 — Placebo, oral, by mouth (Cohort 1 only)
  Arms: Cohort 1
Drug: Placebo Cohort 2 — Placebo, oral, by mouth (Cohort 2 only)
  Arms: Cohort 2
Drug: Placebo for Mirabegron — Placebo for Mirabegron, oral, by mouth (Cohort 3 only)
  Arms: Cohort 3

SUMMARY:
Background:

- Changes in how a person's body burns energy or calories can affect their weight over time. The lowest level of energy the body needs to function is called basal metabolic rate. In the cold, we burn extra energy, even before we start to shiver. This is called non-shivering thermogenesis and it occurs in different types of tissue such as muscle and fat. Researchers want to learn more about this type of energy burning and how it is regulated. They hope this will help treat obesity in the future.

Objectives:

* Sub-study 1: to better understand how non-shivering thermogenesis works.
* Sub-study 2: to measure the effects of anti-obesity drugs on basal metabolic rate.
* Sub-study 3: to better understand the effects of mirabegron, a beta-3 adrenergic receptor agonist, on brown fat activity.

Eligibility:

- Healthy, lean adult males ages 18 to 35.

Design:

* Participants will be screened with medical history, physical exam, blood test, and EKG.
* For sub-studies 1 and 2:

  * Participants will receive one X-ray scan.
  * Each day, all participants will:
* Have height and weight measured, and have urine collected.
* Spend 4 hours in a temperature-controlled room with furniture, toilet area, phone, and computer. They will wear small non-invasive devices to monitor activity, heart rate, temperature, and shivering.
* Walk for 30 minutes.
* For sub-study 3:

  * Participants will receive one DXA scan and up to 4 PET/CT scans and 4 MRIs
  * Each stay, all participants will:
* Have height and weight measured, and have urine collected.
* Spend 6 hours in a temperature-controlled room with furniture, toilet area, phone, and computer. They will wear small non-invasive devices to monitor activity, heart rate, temperature, and shivering.
* Participants will be compensated for their time and participation at the end of the study

DETAILED DESCRIPTION:
The balance between energy expenditure (EE) and energy intake ultimately determines body weight. Resting EE is the major component (60-75%) of total EE in an adult human being. Resting EE dynamically adapts to environmental changes such as ambient temperature. In our on-going study of environmental temperature changes within and around the thermoneutral zone, we observed that healthy young men can increase EE by 17 % of the basal metabolic rate through the process of non-shivering thermogenesis (NST). This capacity for NST is unexpectedly large as compared to prior reports of mild cold-induced thermogenesis (3 to 11%) and suggests that increasing NST could be explored as an intervention to combat obesity.

The aim of this study is to better understand the physiology of NST and to develop improved assays for evaluating the effect of drugs that alter EE. For example, only recently has it been realized that brown adipose tissue (BAT) is functional in adult humans and that white adipose tissue can be converted to brown-adipose-like tissue to increase heat production during cold exposures. Moreover, skeletal muscle likely also plays a role in cold-induced thermogenesis even before overt shivering occurs. It is plausible that the mechanisms governing heat production for NST contribute to regulation of body weight and thus may be contributing to the current obesity epidemic: even small changes in EE, if not compensated by changes in food intake, can have long-term effects on body weight.

This protocol has two phases. The first uses a pharmacologic approach to investigate the mechanism of NST in young healthy lean males. Since the principal physiologic stimulus to BAT (and possibly muscle for NST) is via the sympathetic nervous system (SNS), beta-adrenergic receptors may hold key roles in regulating human EE. We hypothesize that, by careful measurements of NST (at an individually-titrated cool environmental temperature, between 18 21 degrees C vs. at thermoneutrality of 27 degrees C) and using beta-adrenergic drugs that differ in receptor specificity and agonist/antagonist properties, we will gain better understanding of the regulation of human NST.

The second phase of the study focuses on measuring of FDA-approved drugs (such as anti-obesity drugs) potential effect on basal metabolic rate (BMR) under thermoneutral conditions. The rationale is that previous studies of drug effect on EE in humans have not always rigorously enforced the use of thermoneutral conditions, thus may have increased variability and underestimated the effect, contributing to inconclusive findings.

It is envisioned that this study will further our knowledge of the mechanisms that regulate the acute adaptive changes in resting energy expenditure and the effects of drug therapy targeting obesity in humans.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Generally healthy
* Males between the age 18-35 years
* Written informed consent.

EXCLUSION CRITERIA:

* BMI less than 18.5 or greater than 25.0 kg/M(2)
* History of cardiovascular disease such as congestive heart failure, heart block, clinically abnormal EKG as determined by investigators
* History of liver disease or ALT serum level greater than two times the laboratory upper limit of normal
* History of kidney diseases or renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min (MDRD equation)
* History of cancer or bariatric surgery
* History of diabetes mellitus or fasting serum glucose > 126 mg/dL
* History of hypo- or hyper-thyroid or abnormal TSH, except minor deviations deemed to be of no clinical significance by the investigator.
* History of asthma, chronic obstructive pulmonary disease and glaucoma
* Psychological conditions, such as (but not limited to) claustrophobia, clinical depression, bipolar disorders, that would be incompatible with safe and successful participation in this study
* Weight change >5 percent in the past 6 months or a trained athlete
* Blood pressure greater than 140/90 mmHg or current antihypertensive therapy
* Iron deficiency (Hemoglobin <13.7 g/dL and Hematocrit <40.1%)
* History of illicit drug, opioids, or alcohol abuse within the last 5 years; current use of drugs (by history) or alcohol (CAGE greater than or equal to 2) (95)
* Current use of medications/dietary supplements/alternative therapies known to alter energy metabolism
* Current medications that may have interactions with study drugs as determined by the investigators
* History of adverse or allergic reactions to the study drugs
* Daily caffeine intake >500 mg (about 4 cups) and have withdrawal symptoms
* Current smoker or user of tobacco products
* Cannot commit to the schedule of visits to the Clinical Research Center (CRC) as required by the study timeline
* Have had previous radiation exposure within the last year (X-rays, PET scans, etc.) that would exceed research limits (please let us know if you have received radiation for research purposes)
* Have inflexible dietary restrictions
* Any other reason that the investigator thinks would make interpretation of the study results difficult.
* For subjects having an MRD (cOHORT 3), history of pacemaker, metallic heart valves, aneurysm clip, pedicle screws, metallic foreign body in eye, or other metallic implant.
* For subjects receiving mirabegron (Cohort 3), a diagnosis of bladder outlet obstruction or the use of antimuscarinic medications for the treatment of overactive bladder.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available by request to the PI following publication of results
Access Criteria: By request to PI with approved protocol to analyze IPD

REFERENCES:
- [Background] Cannon B, Nedergaard J. Nonshivering thermogenesis and its adequate measurement in metabolic studies. J Exp Biol. 2011 Jan 15;214(Pt 2):242-53. doi: 10.1242/jeb.050989. PMID 21177944
- [Background] van Marken Lichtenbelt WD, Schrauwen P. Implications of nonshivering thermogenesis for energy balance regulation in humans. Am J Physiol Regul Integr Comp Physiol. 2011 Aug;301(2):R285-96. doi: 10.1152/ajpregu.00652.2010. Epub 2011 Apr 13. PMID 21490370
- [Background] Nedergaard J, Bengtsson T, Cannon B. Unexpected evidence for active brown adipose tissue in adult humans. Am J Physiol Endocrinol Metab. 2007 Aug;293(2):E444-52. doi: 10.1152/ajpendo.00691.2006. Epub 2007 May 1. PMID 17473055
- [Derived] Baskin AS, Linderman JD, Brychta RJ, McGehee S, Anflick-Chames E, Cero C, Johnson JW, O'Mara AE, Fletcher LA, Leitner BP, Duckworth CJ, Huang S, Cai H, Garraffo HM, Millo CM, Dieckmann W, Tolstikov V, Chen EY, Gao F, Narain NR, Kiebish MA, Walter PJ, Herscovitch P, Chen KY, Cypess AM. Regulation of Human Adipose Tissue Activation, Gallbladder Size, and Bile Acid Metabolism by a beta3-Adrenergic Receptor Agonist. Diabetes. 2018 Oct;67(10):2113-2125. doi: 10.2337/db18-0462. Epub 2018 Jul 6. PMID 29980535
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0200.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 16 | 18 | 13
Completed | 16 | 17 | 12
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Chamber temperature will be block randomized with low temperature and 27C (Cohort 1 only)
  Within each block, the following five interventions will be repeated:
  Propranolol: Propanolol 160mg, oral, by mouth (Cohort 1 only)
  Pindolol: Pindolol 20mg, oral, by mouth (Cohort 1 only)
  Dantrolene: Dantrolene 100mg, oral, by mouth (Cohort 1 only)
  Magnesium Sulfate: Magnesium Sulfate, infusion, 50 mg/kg bolus followed by maintenance infusion at 2g/h (Cohort 1 only)
  Placebo Cohort 1: Placebo, oral, by mouth (Cohort 1 only)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 16 | 18 | 13 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4.6) | 28.1 (4) | 25.1 (4.6) | 26.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 16 | 18 | 13 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 5 | 15
  White | 9 | 11 | 7 | 27
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Resting Energy Expenditure at Low Temperature
Description: Resting energy expenditure (REE) at a temperature just above the subject's placebo shivering threshold.
Time Frame: Cohort 1: Days 1-17
Population: Cohort 1
Measure: Mean (Standard Deviation); unit: kcal/min
Groups:
- Cohort 1: Chamber temperature will be block randomized with low temperature (Cohort 1 only)
  Within each block, the following five interventions will be repeated:
  Propranolol: Propanolol 160mg, oral, by mouth (Cohort 1 only)
  Pindolol: Pindolol 20mg, oral, by mouth (Cohort 1 only)
  Dantrolene: Dantrolene 100mg, oral, by mouth (Cohort 1 only)
  Magnesium Sulfate: Magnesium Sulfate, infusion, 50 mg/kg bolus followed by maintenance infusion at 2g/h (Cohort 1 only)
  Placebo Cohort 1: Placebo, oral, by mouth (Cohort 1 only)
Arm/Group | Cohort 1
Number analyzed (Participants) | 16
kcal/min
  Placebo Cohort 1 | 1.277 (0.151)
  Propranolol | 1.134 (0.109)
  Dantrolene | 1.300 (0.118)
  Magnesium sulfate: number analyzed (Participants) | 15
  Magnesium sulfate | 1.271 (0.126)
  Pindolol: number analyzed (Participants) | 15
  Pindolol | 1.165 (0.112)

2. Primary Outcome: Resting Energy Expenditure at Low Temperature
Description: Resting energy expenditure (REE) at a temperature just above the subject's placebo shivering threshold.
Time Frame: Cohorts 2: Six one-day overnight inpatient stays over a six to twelve week period.
Population: missed visits due to Covid etc.
Measure: Mean (Standard Deviation); unit: kcal/min
Arm/Group | Cohort 2
Number analyzed (Participants) | 18
kcal/min
  Caffeine: number analyzed (Participants) | 15
  Caffeine | 1.292 (0.123)
  Phentermine: number analyzed (Participants) | 14
  Phentermine | 1.217 (0.116)
  Topiramate: number analyzed (Participants) | 13
  Topiramate | 1.191 (0.122)
  Qsymia: number analyzed (Participants) | 13
  Qsymia | 1.228 (0.122)
  Naltrexone: number analyzed (Participants) | 17
  Naltrexone | 1.185 (0.140)
  Placebo: number analyzed (Participants) | 14
  Placebo | 1.215 (0.109)

3. Primary Outcome: Resting Energy Expenditure at Low Temperature
Description: Resting energy expenditure (REE) at a temperature just above the subject's placebo shivering threshold.
Time Frame: Cohort 3: Four one-day overnight inpatient stays over a 12-week period.
Population: missed visits due to Covid etc.
Measure: Mean (Standard Deviation); unit: kcal/min
Arm/Group | Cohort 3
Number analyzed (Participants) | 12
kcal/min
  Placebo for Mirabegron: number analyzed (Participants) | 11
  Placebo for Mirabegron | 1.25 (0.39)
  Mirabegron 50mg | 1.31 (0.19)
  Mirabegron 200mg | 1.37 (0.19)

4. Primary Outcome: Basal Metabolic Rate
Description: Basal metabolic rate (BMR) is the resting energy expenditure (REE) at thermoneutrality (27c).
Time Frame: Cohort 1: Days 1-17
Population: Cohort 1
Measure: Mean (Standard Deviation); unit: kcal/min
Groups:
- Cohort 1: Chamber temperature will be block randomized with 27C (Cohort 1 only)
  Within each block, the following five interventions will be repeated:
  Propranolol: Propanolol 160mg, oral, by mouth (Cohort 1 only)
  Pindolol: Pindolol 20mg, oral, by mouth (Cohort 1 only)
  Dantrolene: Dantrolene 100mg, oral, by mouth (Cohort 1 only)
  Magnesium Sulfate: Magnesium Sulfate, infusion, 50 mg/kg bolus followed by maintenance infusion at 2g/h (Cohort 1 only)
  Placebo Cohort 1: Placebo, oral, by mouth (Cohort 1 only)
Arm/Group | Cohort 1
Number analyzed (Participants) | 16
kcal/min
  Placebo Cohort 1 | 1.153 (0.098)
  Propranolol | 1.053 (0.099)
  Dantrolene | 1.143 (0.105)
  Magnesium sulfate | 1.108 (0.124)
  Pindolol | 1.116 (0.109)

5. Primary Outcome: Brown Adipose Tissue Activity (Cohort 3 Only)
Description: Brown adipose tissue (BAT) activity is a quantification of tissue volume and metabolic activity per unit volume.
Time Frame: Cohort 3: Four one-day overnight inpatient stays over a 12-week period.
Population: missed visits due to Covid etc.
Measure: Mean (Standard Deviation); unit: mL*SUVmean*g/mL
Arm/Group | Cohort 3
Number analyzed (Participants) | 12
mL*SUVmean*g/mL
  Placebo for Mirabegron: number analyzed (Participants) | 11
  Placebo for Mirabegron | 0.1 (0.2)
  Mirabegron 50 mg | 215.3 (446.2)
  Mirabegron 200mg | 554.3 (903.4)

ADVERSE EVENTS:
Time Frame: Twelve weeks
Groups:
- Cohort 1 Low Temperature : Placebo; Cohort 1 Low Temperature : Proprannolol; Cohort 1 Low Temperature : Dantrolene; Cohort 1 Low Temperature : Magnesium; Cohort 1 Low Temperature : Pindolol; Cohort 1 High Temperature : Placebo; Cohort 1 High Temperature : Proprannolol; Cohort 1 High Temperature : Dantrolene; Cohort 1 High Temperature : Magnesium; Cohort 1 High Temperature : Pindolol: Chamber temperature will be block randomized with low temperature and 27C (Cohort 1 only)
  Within each block, the following five interventions will be repeated:
  Propranolol: Propanolol 160mg, oral, by mouth (Cohort 1 only)
  Pindolol: Pindolol 20mg, oral, by mouth (Cohort 1 only)
  Dantrolene: Dantrolene 100mg, oral, by mouth (Cohort 1 only)
  Magnesium Sulfate: Magnesium Sulfate, infusion, 50 mg/kg bolus followed by maintenance infusion at 2g/h (Cohort 1 only)
  Placebo Cohort 1: Placebo, oral, by mouth (Cohort 1 only)
- Cohort 2 : Placebo; Cohort 2 : Caffeine; Cohort 2 : Naltrexone; Cohort 2 : Qsymia; Cohort 2 : Topiramate; Cohort 2 : Phentermine: Interventions, in random order, will be administered during one of the six one-day stays
  Caffeine: Caffeine 200mg, oral, by mouth (Cohort 2 only)
  Qsymia: Qsymia (topiramate 92mg CR, phentermine 15mg PO), oral, by mouth (Cohort 2 only)
  Topiramate: Topiramate 200mg, oral, by mouth (Cohort 2 only)
  Phentermine: Phentermine 37.5mg, oral, by mouth (Cohort 2 only)
  Naltrexone: Naltrexone 100mg, oral, by mouth (Cohort 2 only)
  Placebo Cohort 2: Placebo, oral, by mouth (Cohort 2 only)
- Cohort 3 : Placebo; Cohort 3 : Mirabegron 50mg; Cohort 3 : Mirabegron 200mg: Interventions, in random order, will be administered during one of the four overnight inpatient stays
  Mirabegron 50mg: Mirabegron 50mg, oral, by mouth (Cohort 3 only)
  Mirabegron 200mg: Mirabegron 200mg, oral, by mouth (Cohort 3 only)
  Placebo for Mirabegron: Placebo for Mirabegron, oral, by mouth (Cohort 3 only)
Arm/Group | Cohort 1 Low Temperature : Placebo | Cohort 1 Low Temperature : Proprannolol | Cohort 1 Low Temperature : Dantrolene | Cohort 1 Low Temperature : Magnesium | Cohort 1 Low Temperature : Pindolol | Cohort 1 High Temperature : Placebo | Cohort 1 High Temperature : Proprannolol | Cohort 1 High Temperature : Dantrolene | Cohort 1 High Temperature : Magnesium | Cohort 1 High Temperature : Pindolol | Cohort 2 : Placebo | Cohort 2 : Caffeine | Cohort 2 : Naltrexone | Cohort 2 : Qsymia | Cohort 2 : Topiramate | Cohort 2 : Phentermine | Cohort 3 : Placebo | Cohort 3 : Mirabegron 50mg | Cohort 3 : Mirabegron 200mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 1/16 | 0/16 | 0/16 | 1/16 | 0/16 | 0/16 | 1/16 | 0/18 | 0/18 | 5/18 | 2/18 | 5/18 | 2/18 | 1/13 | 1/13 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Low Temperature : Placebo (N=16) | Cohort 1 Low Temperature : Proprannolol (N=16) | Cohort 1 Low Temperature : Dantrolene (N=16) | Cohort 1 Low Temperature : Magnesium (N=16) | Cohort 1 Low Temperature : Pindolol (N=16) | Cohort 1 High Temperature : Placebo (N=16) | Cohort 1 High Temperature : Proprannolol (N=16) | Cohort 1 High Temperature : Dantrolene (N=16) | Cohort 1 High Temperature : Magnesium (N=16) | Cohort 1 High Temperature : Pindolol (N=16) | Cohort 2 : Placebo (N=18) | Cohort 2 : Caffeine (N=18) | Cohort 2 : Naltrexone (N=18) | Cohort 2 : Qsymia (N=18) | Cohort 2 : Topiramate (N=18) | Cohort 2 : Phentermine (N=18) | Cohort 3 : Placebo (N=13) | Cohort 3 : Mirabegron 50mg (N=13) | Cohort 3 : Mirabegron 200mg (N=13)
Asymptomatic non-sustained ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter-related asymptomatic uncomplicated right upper extremity superficial venous thrombophlebiti (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncopal episode, likely vasovagal response (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Right lower lung subcentimeter pleural based nodular density (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Incidental PET CT- Right upper lung subcentimeter nodule associated with hypermetabolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incidental PET CT- Nonspecific subpleural nodules (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0
Presyncopal episode, likely vasovagal response (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Feels foggy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 0 | 0 | 0 | 0
Drowsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Feels edgy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Fatigue (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT01950520/Prot_SAP_000.pdf